CLINICAL TRIAL: NCT03464136
Title: A Phase 3b, Multicenter, Randomized, Blinded, Active-Controlled Study to Compare the Efficacy and Safety of Ustekinumab to That of Adalimumab in the Treatment of Biologic Naïve Subjects With Moderately-to-Severely Active Crohn's Disease
Brief Title: Safety and Efficacy of Adalimumab Versus Ustekinumab for One Year
Acronym: SEAVUE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR108449; 2017-004209-41 (EudraCT Number); CNTO1275CRD3007 (Other: Janssen Scientific Affairs, LLC)
Record Dates: First submitted 2018-03-07; First posted 2018-03-13 (Actual); Results first posted 2022-01-11 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Ustekinumab; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Ustekinumab) (Experimental): Participants will receive intravenous (IV) infusion of ustekinumab (approximately 6 milligram/kilogram [mg/kg]) and 4 subcutaneous (SC) injections of placebo for adalimumab at Week 0, followed by 2 SC injections of placebo at Week 2. From Week 4 to Week 56, participants will self-administer one SC injection of ustekinumab 90 milligram (mg) every 8 weeks (q8w) starting at Week 8 and placebo adalimumab at the other designated every 2 weeks (q2w) dosing intervals.
  Interventions: Biological: Placebo for Ustekinumab; Biological: Ustekinumab (6 mg/kg); Biological: Ustekinumab (90 mg)
- Group 2 (Adalimumab) (Active Comparator): Participants will receive IV infusion of placebo for ustekinumab and 4 SC injections of adalimumab (each 40 mg, total dose 160 mg) at Week 0, followed by 2 SC injections of adalimumab (each 40 mg, total dose 80 mg) at Week 2. From Week 4 to Week 56, participants will self-administer 1 SC injection of adalimumab 40 mg q2w.
  Interventions: Biological: Placebo for Adalimumab; Biological: Adalimumab (40 mg)

INTERVENTIONS:
Biological: Placebo for Ustekinumab — Participants will receive placebo as SC injection to blind adalimumab.
  Arms: Group 1 (Ustekinumab)
Biological: Placebo for Adalimumab — Participants will receive placebo as IV infusion to blind ustekinumab.
  Arms: Group 2 (Adalimumab)
Biological: Ustekinumab (6 mg/kg) — Participants will receive ustekinumab 6 mg/kg (weight based dosing) as IV infusion.
  Other Names: Stelara
  Arms: Group 1 (Ustekinumab)
Biological: Ustekinumab (90 mg) — Participants will self-administer SC injection of ustekinumab 90 mg.
  Other Names: Stelara
  Arms: Group 1 (Ustekinumab)
Biological: Adalimumab (40 mg) — Participants will self-administer multiple SC injections of adalimumab (each 40 mg) and will receive total dose of 160 mg at Week 0, 80 mg at Week 2, and 40 mg q2w from Week 4 to 56.
  Other Names: Humira
  Arms: Group 2 (Adalimumab)

SUMMARY:
The purpose of this study is to compare the efficacy of treatment with ustekinumab or adalimumab in biologic naive participants with moderately-to-severely active Crohn's disease (CD) who have previously failed or were intolerant to conventional therapy (corticosteroids and/or immunomodulators, such as azathioprine, 6-mercaptopurine, or methotrexate), as measured by clinical remission at one year.

DETAILED DESCRIPTION:
This study compares the safety and efficacy of ustekinumab versus adalimumab. It will consist of screening (within 1- 5 weeks prior to Week 0), treatment phase (Weeks 0 to 52), and follow-up phase (up to Week 76). The primary hypothesis is that ustekinumab is superior to adalimumab as measured by clinical remission after one year of treatment. Study assessments will include Crohn's disease activity index (CDAI), video ileocolonoscopy; CD-related healthcare utilization; patient-reported outcomes (PROs); laboratory evaluations; biomarkers; review of concomitant medications and adverse events (AEs); and evaluation of serum concentrations of study agent as well as development of antibodies to study agent. All participants will randomly be assigned to receive either ustekinumab or adalimumab. No participants will be treated with placebo only.

ELIGIBILITY:
Inclusion Criteria:

* Has Crohn's Disease (CD) or fistulizing CD of at least 3 months' duration, with colitis, ileitis, or ileocolitis, confirmed at some time in the past by radiography, histology, and/or endoscopy
* Has moderately-to-severely active CD with a baseline Crohn's disease activity index (CDAI) score of greater than or equal to (>=) 220 and less than or equal to (<=) 450
* Has one or more ulceration on screening ileocolonoscopy (which by definition, would result in an Simple Endoscopic Score for Crohn's Disease [SES-CD] of at least 3)
* Has failed or was intolerant to conventional therapy (corticosteroids, azathioprine [AZA], 6-mercaptopurine [6-MP] and/or methotrexate [MTX]) at adequate doses or is corticosteroid dependent
* Has not previously received an approved biologic for Crohn's Disease (i.e., infliximab, adalimumab, certolizumab pegol, ustekinumab, natalizumab, vedolizumab or approved biosimilars of these agents)
* Participants on oral corticosteroids (e.g., prednisone, budesonide) at a prednisone-equivalent dose of <=40 or milligram/day (mg/day) or <=9 mg/day of budesonide are budesonide <=9 mg/day are permitted if doses are stable for 3 weeks prior to baseline
* Participants on AZA, 6-MP, or MTX at screening (or recently prior), must discontinue these medications at least 3 weeks prior to baseline

Exclusion Criteria:

* Has complications of CD that are likely to require surgery or would confound the ability to assess the effect of ustekinumab or adalimumab treatment using the CDAI, such as: active stoma; short-gut syndrome and severe or symptomatic strictures or stenosis
* Currently has, or is suspected to have, an abscess. Recent cutaneous and perianal abscesses are not exclusionary if drained and adequately treated at least 3 weeks prior to baseline, or 8 weeks prior for intra-abdominal abscesses, if there is no anticipated need for any further surgery. Participants with active fistulas may be included if there is no anticipation of a need for surgery and there are currently no abscesses present
* Has had any kind of bowel resection within 6 months prior to baseline or other intra-abdominal surgery or a hospital admission for bowel obstruction within 3 months prior to baseline
* Has a stool culture or other examination positive for an enteric pathogen, including Clostridium difficile toxin, in the last 4 months unless a repeat examination is negative and there are no signs of ongoing infection with that pathogen
* Has received a Bacillus Calmette-Guerin (BCG) vaccination within 12 months or any other live bacterial or live viral vaccination within 2 weeks of baseline
* Has a history of, or ongoing, chronic or recurrent infectious disease, including but not limited to, chronic renal infection, chronic chest infection, recurrent urinary tract infection (eg, recurrent pyelonephritis or chronic nonremitting cystitis), or infected skin wounds or ulcers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Janssen Scientific Affairs, LLC
Locations (182):
- United States (67):
  - Alabama Medical Group, Mobile, Alabama
  - Precision Research Institute, San Diego, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Gastro Associates of Fairfield County PC, Bridgeport, Connecticut
  - Western Connecticut Health Network/Danbury Hospital, Danbury, Connecticut
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Gastro Florida, Clearwater, Florida
  - Florida Research Network, LLC, Gainesville, Florida
  - Florida Center For Gastroenterology, Largo, Florida
  - Center for Advanced Gastroenterology, Maitland, Florida
  - Gastroenterology Group Of Naples, Naples, Florida
  - Advanced Medical Research Center, Port Orange, Florida
  - Apex Clinical Research, Tampa, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Atlanta Gastroenterology Specialists, PC, Suwanee, Georgia
  - Grand Teton Research Group, PLLC, Idaho Falls, Idaho
  - Health Science Research Center, Pratt, Kansas
  - Tri-State Gastroenterology Assoc, Crestview Hills, Kentucky
  - Gastroenterology Associates Of Hazard, Hazard, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Texas Digestive Disease Consultants, Baton Rouge, Louisiana
  - CroNOLA, LLC, Houma, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Huron Gastroenterology Associates Center for Digestive Care, Ypsilanti, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Saint Louis University Hospital, St Louis, Missouri
  - Mercy Clinic East Community, St Louis, Missouri
  - Saratoga Schenectady Gastroenterology Associates, Burnt Hills, New York
  - NYU Langone Long Island Clinical Research Associates, Great Neck, New York
  - Weill Cornell Medical College, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Columbia University Medical Center, New York, New York
  - Premier Medical Group Of The Hudson Valley, Pc, Poughkeepsie, New York
  - University of Rochester Medical Center, Rochester, New York
  - Digestive Health Partners, Asheville, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Hospital Medical Center, Raleigh, North Carolina
  - Wilmington Gastroenterology Associates, Wilmington, North Carolina
  - Fargo Gastroenterology Clinic, PC, Fargo, North Dakota
  - Northshore Gastroenterology Research, LLC, Beachwood, Ohio
  - TriHealth Digestive Institute, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Ohio State University Hospital, Columbus, Ohio
  - Dayton Gastroenterology, Inc, Dayton, Ohio
  - Great Lakes Gastroenterology Research, LLC, Mentor, Ohio
  - Digestive Disease Specialists Inc, Oklahoma City, Oklahoma
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Allegheny-Singer Research Institute, Pittsburgh, Pennsylvania
  - Gastroenterology Associates P.A., Greenville, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Aztec Clinical Research, Inc., Channelview, Texas
  - DHAT Research Institute, Garland, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Texas at Houston Medical School, Houston, Texas
  - Gastroenterology Research of America, LLC, San Antonio, Texas
  - Texas Digestive Disease Consultants, Southlake, Texas
  - Tyler Research Institute, LLC, Tyler, Texas
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
  - Verity Research, Inc, Fairfax, Virginia
  - Gastroenterology Associates of Central Virginia, Lynchburg, Virginia
  - Digestive And Liver Disease Specialists, Norfolk, Virginia
  - McGuire VAMC, Richmond, Virginia
  - Virginia Gastroenterology Institute, Suffolk, Virginia
  - Washington Gastroenterology, PLLC, Bellevue, Washington
  - Washington Gastroenterology, PLLC, Tacoma, Washington
- Australia (5):
  - Monash Health, Monash Medical Centre, Clayton
  - Alfred Hospital, Melbourne
  - Mater Hospital Brisbane Inflammatory Bowel Diseases, South Brisbane
  - St John of God Subiaco Hospital, Subiaco
  - The Queen Elizabeth Hospital, Woodville South
- Belgium (3):
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
  - CHwapi, Tournai
- Brazil (8):
  - Hospital Das Clinicas Da Ufmg, Belo Horizonte - MG
  - Inst Goiano Gastroenterologia e Endoscopia Digest Ltda - Clinica de Gastro, Goiânia
  - Endogastro Clínica de Gastroenterologia e Endoscopia Digestiva Lida, Juiz de Fora
  - Hospital das Clinicas de Porto Alegre, Porto Alegre
  - Hospital Das Clinicas Da Faculdade De Medicina De RPUSP HCRP, Ribeirão Preto
  - Universidade Federal do Rio de Janeiro - Faculdade de Medicina, Rio de Janeiro
  - Hospital Copa D'Or, Rio de Janeiro
  - Fundacao do ABC Centro Universitario FMABC, Santo André
- Bulgaria (4):
  - UMHAT 'Dr. Georgi Stranski', EAD, Pleven
  - MHAT Rousse, Rousse
  - 2-nd MHAT, Sofia
  - Diagnostic Consulting Center Mladost - M Varna, Varna
- Canada (5):
  - University of Calgary, Calgary, Alberta
  - McMaster University, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - CISSS de la Monteregie Centre, Greenfield Park, Quebec
  - CMIIM, Centre médical L'Enjeu, Mount Royal, Quebec
- Czechia (5):
  - Fakultní nemocnice u sv. Anny v Brn, Brno
  - Nemocnice Horovice, a.s., Hořovice
  - Hepato-gastroenterologie HK, s.r.o., Hradec Králové
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - ISCARE a.s., Prague
- France (6):
  - CHU Amiens, Amiens
  - CHRU Montpellier - Hopital Saint-Eloi, Montpellier
  - Hotel Dieu, Nantes
  - Hopital Saint Louis, Paris
  - CHU Saint Etienne, Saint-Priest-en-Jarez
  - Clinique Ambroise Pare, Toulouse
- Germany (4):
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - Asklepios Westklinikum, Hamburg
  - Uniklinikum Heidelberg, Heidelberg
  - MVZ Portal10, Münster
- Hungary (6):
  - Réthy Pál Kórház - Rendelőintézet, Békéscsaba
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Semmelweis Egyetem, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Borsod-Abauj-Zemplen Megyei Korhaz es Egyetemi Oktato Korhaz, Miskolc
  - Markusovszky Egyetemi Oktatokorhaz, Szombathely
- Italy (11):
  - Policlinico Sant'Orsola Malpighi, Bologna
  - AOU Policlinico G.Martino, Messina
  - ASST Fatebenefratelli Sacco, Milan
  - Azienda Ospedaliera di Padova, Padua
  - Ospedale Villa Sofia-Cervello, Palermo
  - Azienda Ospedaliera G.Salvini Ospedale di Rho, Rho
  - Azienda Ospedaliera Universitaria 'Policlinico Tor Vergata', Roma
  - Azienda Complesso Ospedaliero San Filippo Neri, Roma
  - Fondazione Policlinico Gemelli Università Cattolica, Roma
  - Istituto Clinico Humanitas, Rozzano
  - AO Ordine Mauriziano, Torino
- Netherlands (7):
  - VUMC Amsterdam, Amsterdam
  - Rijnstate Ziekenhuis, Arnhem
  - UMCG, Groningen
  - Leiden University Medical Center, Leiden
  - Radboudumc, Nijmegen
  - Sint Franciscus Gasthuis, Rotterdam
  - Ikazia Ziekenhuis, Rotterdam
- Poland (13):
  - Gastromed Kralisz Romatowski Stachurska Sp. j., Bialystok
  - Synexus Polska Sp z o o, Gdansk
  - Centrum Medyczne Plejady, Krakow
  - Centrum Medyczne Pratia Poznan, Krakow
  - Uniwersytecki Szpital Kliniczny nr 1 im. N. Barlickiego, Lodz
  - Samodzielny Publiczny Szpital Kliniczny Nr 4 w Lublinie Oddzial Gastroenterologii, Lublin
  - Centrum Medyczne Medyk, Rzeszów
  - Endoskopia Sp z o o z siedziba w Sopocie, Sopot
  - Centralny Szpital Kliniczny MSWiA w Warszawie, Warsaw
  - Niepubliczny Zaklad Opieki Zdrowotnej Vivamed Jadwiga Miecz, Warsaw
  - Gabinety Lekarskie Bodyclinic, Warsaw
  - Melita Medical Sp. z o.o., Wroclaw
  - ETG Zamosc, Zamość
- Russia (8):
  - Irkutsk State Medical Academy of Postgraduate Education, Irkutsk
  - GU Moscow Regional Research Clinical Institute n.a. M.F.Vla, Moscva
  - Rostov State Medical University, Rostov-on-Don
  - Elizavetinskaya hospital, Saint Petersburg
  - City Clinical Hospital #31, Saint Petersburg
  - GBUZ Respublican Clinical Hospital n.a. GG Kuvatova, Ufa
  - City Clinical Hospital # 21, Ufa
  - OOO MO New Hospital, Yekaterinburg
- Serbia (6):
  - Clinical Hospital Center Zemun, Belgrade
  - Clinical Hospital Center Zvezdara, Belgrade
  - University Clinical Center Kragujevac, Kragujevac
  - University Clinical Center NIS, Niš
  - Clinical Center of Vojvodina, Vojvodina
  - Clinical Hospital Center Bezanijska Kosa, Zemun
- South Korea (7):
  - Yeungnam University Hospital, Daegu
  - The Catholic university of Korea, St. Vincent's Hospital, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
- Spain (10):
  - Hosp. Del Mar, Barcelona
  - Hosp. de La Santa Creu I Sant Pau, Barcelona
  - Hosp. Univ. Dr. Josep Trueta, Girona
  - Hosp. Univ. Central de Asturias, Oviedo
  - Corporacio Sanitari Parc Tauli, Sabadell
  - Hosp Clinico Univ de Salamanca, Salamanca
  - Hosp. Univ. Marques de Valdecilla, Santander
  - Hosp. Virgen Macarena, Seville
  - Hosp. Univ. Rio Hortega, Valladolid
  - Hosp. Univ. Miguel Servet, Zaragoza
- United Kingdom (7):
  - Royal United Hospital, Bath
  - Pennine Acute Hospitals-Fairfield General Hospital, Bury
  - Kingston Hospital, Kingston upon Thames
  - Guy's and St Thomas' Hospital, London
  - St George's Hospital, London
  - Southampton University Hospitals NHS Trust, Southampton
  - Musgrove Park Hospital, Taunton

REFERENCES:
- [Derived] Venkat S, Zeeman M, Hart A, Bhagat S, Galbraith DA, Hoops T, Ufberg PJ, Izanec J, Freeman TC, Mcrae B, Shinzaki S, Jairath V, Panaccione R, Sands BE, Branigan P. Serum protein profiles differ with adalimumab and ustekinumab treatment in moderately to severely active Crohn's disease. J Crohns Colitis. 2025 Dec 5;19(11):jjaf197. doi: 10.1093/ecco-jcc/jjaf197. PMID 41258994
- [Derived] Hasskamp J, Meinhardt C, Timmer A. Anti-IL-12/23p40 antibodies for induction of remission in Crohn's disease. Cochrane Database Syst Rev. 2025 May 13;5(5):CD007572. doi: 10.1002/14651858.CD007572.pub4. PMID 40357993
- [Derived] Sands BE, Irving PM, Hoops T, Izanec JL, Gao LL, Gasink C, Greenspan A, Allez M, Danese S, Hanauer SB, Jairath V, Kuehbacher T, Lewis JD, Loftus EV Jr, Mihaly E, Panaccione R, Scherl E, Shchukina OB, Sandborn WJ; SEAVUE Study Group. Ustekinumab versus adalimumab for induction and maintenance therapy in biologic-naive patients with moderately to severely active Crohn's disease: a multicentre, randomised, double-blind, parallel-group, phase 3b trial. Lancet. 2022 Jun 11;399(10342):2200-2211. doi: 10.1016/S0140-6736(22)00688-2. PMID 35691323

RESULTS

PARTICIPANT FLOW:
Groups:
- Adalimumab: Participants received intravenous (IV) infusion of placebo for ustekinumab and 4 subcutaneous (SC) injections of adalimumab (each 40 milligrams [mg], total dose 160 mg) at Week 0, followed by 2 SC injections of adalimumab (each 40 mg, total dose 80 mg) at Week 2. From Week 4 to Week 56, participants self-administered 1 SC injection of adalimumab 40 mg every 2 weeks (q2w).
- Ustekinumab: Participants received IV infusion of ustekinumab (approximately 6 milligram/kilogram [mg/kg]) and 4 SC injections of placebo for adalimumab at Week 0, followed by 2 SC injections of placebo at Week 2. From Week 4 to Week 56, participants self-administered one SC injection of ustekinumab 90 mg every 8 weeks (q8w) starting at Week 8 and placebo adalimumab at the other designated q2w dosing intervals.
Period: Overall Study
Arm/Group | Adalimumab | Ustekinumab
Started | 195 | 191
Completed | 165 | 166
Not Completed | 30 | 25
Not completed — Lost to Follow-up | 5 | 8
Not completed — Withdrawal by Subject | 16 | 13
Not completed — Death | 1 | 0
Not completed — Other | 8 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adalimumab | Ustekinumab | Total
Number analyzed (Participants) | 195 | 191 | 386
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (12.99) | 37 (13.23) | 37.2 (13.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 101 | 201
  Male | 95 | 90 | 185
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 14 | 28
  Not Hispanic or Latino | 178 | 173 | 351
  Unknown or Not Reported | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 11 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 8 | 15
  White | 181 | 164 | 345
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 1 | 6 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 5 | 2 | 7
  Belgium | 2 | 3 | 5
  Brazil | 9 | 14 | 23
  Bulgaria | 5 | 1 | 6
  Canada | 7 | 7 | 14
  Czech Republic | 14 | 8 | 22
  France | 3 | 8 | 11
  Germany | 0 | 1 | 1
  Hungary | 16 | 13 | 29
  Italy | 11 | 10 | 21
  Netherlands | 2 | 5 | 7
  Poland | 34 | 26 | 60
  Republic of Korea | 3 | 8 | 11
  Russia | 27 | 20 | 47
  Serbia | 10 | 2 | 12
  Spain | 4 | 14 | 18
  United Kingdom | 12 | 13 | 25
  United States of America | 31 | 36 | 67

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Remission at Week 52
Description: Percentage of participants with clinical remission at Week 52 were assessed. Clinical remission was defined as a Crohn's Disease Activity Index (CDAI) score of less than (<) 150 points (in general, CDAI score ranges from 0 to approximately 600; higher score indicates higher disease activities). The CDAI score is used to quantify the symptoms of participants with Crohn's Disease. A decrease in CDAI over time indicates improvement in disease activity.
Time Frame: Week 52
Population: Full analysis set (FAS) which was defined as all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab | Ustekinumab
Number analyzed (Participants) | 195 | 191
percentage of participants | 61.0 | 64.9

2. Secondary Outcome: Percentage of Participants With Corticosteroid-free Remission at Week 52
Description: Percentage of participants with Corticosteroid-free remission at Week 52 were assessed. Corticosteroid-free remission was defined as CDAI score <150 points at Week 52 and not taking any corticosteroids for at least 30 days prior to Week 52. The CDAI score is used to quantify the symptoms of participants with Crohn's Disease. CDAI score ranges from 0 to approximately 600; higher score indicates higher disease activities. A decrease in CDAI over time indicates improvement in disease activity.
Time Frame: Week 52
Population: FAS which was defined as all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab | Ustekinumab
Number analyzed (Participants) | 195 | 191
percentage of participants | 57.4 | 60.7

3. Secondary Outcome: Percentage of Participants With Clinical Response at Week 52
Description: Percentage of participants with clinical response at Week 52 were assessed. Clinical response at Week 52 was defined as a reduction from baseline in the CDAI score of greater than or equal (>=) 100 points. The CDAI score is used to quantify the symptoms of participants with Crohn's Disease. CDAI score ranges from 0 to approximately 600; higher score indicates higher disease activities. A decrease in CDAI over time indicates improvement in disease activity.
Time Frame: Week 52
Population: FAS which was defined as all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab | Ustekinumab
Number analyzed (Participants) | 195 | 191
percentage of participants | 66.2 | 72.3

4. Secondary Outcome: Percentage of Participants in Patient Reported Outcome (PRO)-2 Symptom Remission at Week 52
Description: PRO2 evaluated 2 patient-reported symptoms: the frequency of liquid or soft stools (total number of soft/liquid stools in the last 7 days) and abdominal pain (on a 4-point scale where 0 = none, 1 = mild, 2 = moderate, 3 = severe). A weekly score was calculated for the liquid or soft stool frequency and a separate weekly score was calculated for abdominal pain, in each case based on daily symptom reporting. PRO-2 symptom remission was defined as an abdominal pain (AP) mean daily score at or below 1 and also stool frequency (SF) mean daily score at or below 3, that is, AP <=1 and SF <=3. PRO2 is a composite index consisting of weighted scoring of both variables. PRO-2 scores range from 0 to no upper limit with higher scores indicating more severe disease.
Time Frame: Week 52
Population: FAS which was defined as all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab | Ustekinumab
Number analyzed (Participants) | 195 | 191
percentage of participants | 55.4 | 56.5

5. Secondary Outcome: Percentage of Participants With Clinical Remission at Week 16
Description: Percentage of participants with clinical remission (defined as CDAI <150 points) at Week 16 were assessed. Clinical remission was defined as a CDAI score of < 150 points (in general, CDAI score ranges from 0 to approximately 600; higher score indicates higher disease activities). The CDAI score is used to quantify the symptoms of participants with Crohn's Disease. A decrease in CDAI over time indicates improvement in disease activity.
Time Frame: Week 16
Population: FAS which was defined as all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab | Ustekinumab
Number analyzed (Participants) | 195 | 191
percentage of participants | 60 | 57.1

6. Secondary Outcome: Percentage of Participants With Endoscopic Remission at Week 52
Description: Percentage of participants with endoscopic remission at Week 52 were assessed. Endoscopic remission was defined as Simple Endoscopic Score for Crohn's Disease (SES-CD) score less than or equal to (<=) 3, or SES-CD =0 for participants who entered the study with a SES-CD =3 at Week 52. The SES-CD evaluates 4 endoscopic variables (ulcer size, proportion of the surface area that is ulcerated, proportion of the surface area affected, and stenosis) each rated from 0 (best) to 3 (worst) in 5 segments evaluated during ileocolonoscopy (ileum, right colon, transverse colon, left colon, and rectum). The score for each endoscopic variable is the sum of values obtained for each segment. The SES-CD total is the sum of the 4 endoscopic variable scores from 0 to 56, where higher scores indicate more severe disease.
Time Frame: Week 52
Population: FAS among participants with SES-CD Score >=3 at Baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab | Ustekinumab
Number analyzed (Participants) | 179 | 179
percentage of participants | 30.7 | 28.5

7. Secondary Outcome: Percentage of Participants With Clinical Remission Through Week 52
Description: Percentage of participants with clinical remission at each postbaseline visit through Week 52 were reported. Clinical remission was defined as a CDAI score of <150 points (in general, CDAI score ranges from 0 to approximately 600; higher score indicates higher disease activities). The CDAI score is used to quantify the symptoms of participants with Crohn's Disease. A decrease in CDAI over time indicates improvement in disease activity.
Time Frame: Weeks 2, 8, 16, 24, 32, 40, 48, and 52
Population: FAS which was defined as all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab | Ustekinumab
Number analyzed (Participants) | 195 | 191
percentage of participants
  Week 2 | 28.7 | 23.0
  Week 8 | 47.7 | 50.3
  Week 16 | 60.0 | 57.1
  Week 24 | 66.2 | 57.6
  Week 32 | 65.1 | 59.7
  Week 40 | 60.5 | 64.9
  Week 48 | 59.0 | 62.8
  Week 52 | 61.0 | 64.9

8. Secondary Outcome: Percentage of Participants With Clinical Response Through Week 52
Description: Percentage of participants with clinical response at each postbaseline visit through Week 52 were reported. Clinical response through Week 52 was defined as a reduction from baseline in the CDAI score of >=100 points. The CDAI score is used to quantify the symptoms of participants with Crohn's Disease. CDAI score ranges from 0 to approximately 600; higher score indicates higher disease activities. A decrease in CDAI over time indicates improvement in disease activity.
Time Frame: Weeks 2, 8, 16, 24, 32, 40, 48, and 52
Population: FAS which was defined as all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab | Ustekinumab
Number analyzed (Participants) | 195 | 191
percentage of participants
  Week 2 | 46.2 | 38.2
  Week 8 | 66.2 | 68.1
  Week 16 | 72.3 | 73.3
  Week 24 | 76.4 | 70.7
  Week 32 | 74.9 | 71.2
  Week 40 | 69.2 | 74.3
  Week 48 | 66.7 | 69.1
  Week 52 | 66.2 | 72.3

9. Secondary Outcome: Percentage of Participants With Durable Clinical Response at Week 52
Description: Percentage of participants with durable clinical response at Week 52 were reported. Durable clinical response was defined as CDAI score decreased at least 100 from baseline or CDAI <150 at Week 52 and was >= 80% of all visits between Week 16 and Week 52. The CDAI score is used to quantify the symptoms of participants with Crohn's Disease. CDAI score ranges from 0 to approximately 600; higher score indicates higher disease activities. A decrease in CDAI over time indicates improvement in disease activity.
Time Frame: Week 52
Population: FAS which was defined as all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab | Ustekinumab
Number analyzed (Participants) | 195 | 191
percentage of participants | 60.5 | 65.4

10. Secondary Outcome: Percentage of Participants With Durable Clinical Remission at Week 52
Description: Percentage of participants with durable clinical remission at Week 52 were reported. Clinical remission was defined as CDAI score <150 at Week 52 and was >= 80% of all visits between Week 16 and Week 52. The CDAI score is used to quantify the symptoms of participants with Crohn's Disease. CDAI score ranges from 0 to approximately 600; higher score indicates higher disease activities. A decrease in CDAI over time indicates improvement in disease activity.
Time Frame: Week 52
Population: FAS which was defined as all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab | Ustekinumab
Number analyzed (Participants) | 195 | 191
percentage of participants | 51.8 | 50.8

11. Secondary Outcome: Percentage of Participants With Abdominal Pain (AP) Improvement Through Week 52
Description: Percentage of participants with AP improvement through Week 52 were reported. AP improvement was defined as at least 1 point or greater improvement in mean daily CDAI AP score (ranges from 0 to 3 where higher score indicates severity of pain) from baseline, or a mean score of zero among participants with mean AP>0 at baseline, compared at each visit through Week 52.
Time Frame: Weeks 2, 8, 16, 24, 32, 40, 48, and 52
Population: FAS among participants with mean daily AP Score >0 at Baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab | Ustekinumab
Number analyzed (Participants) | 194 | 191
percentage of participants
  Week 2 | 29.9 | 23.0
  Week 8 | 54.1 | 53.9
  Week 16 | 62.9 | 59.2
  Week 24 | 66.5 | 61.8
  Week 32 | 63.9 | 63.9
  Week 40 | 60.3 | 63.9
  Week 48 | 61.9 | 61.8
  Week 52 | 62.4 | 64.9

12. Secondary Outcome: Percentage of Participants With Reduction in Frequency of Diarrhea Through Week 52
Description: Number of participants with reduction in frequency of diarrhea were reported. Reduction in frequency of diarrhea was defined as a reduction of at least 3 (or a mean number <1) in SF (that is, mean daily number of liquid or very soft stools from CDAI score [ranges from 0 to 3 where higher score indicates severity of pain] in the week prior to the visit) from baseline, among subjects with mean SF >1 at baseline, compared at each visit through Week 52.
Time Frame: Weeks 2, 8, 16, 24, 32, 40, 48, and 52
Population: FAS among participants with mean daily stool frequency >1 at Baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab | Ustekinumab
Number analyzed (Participants) | 186 | 179
percentage of participants
  Week 2 | 33.3 | 30.7
  Week 8 | 52.7 | 60.3
  Week 16 | 53.8 | 60.9
  Week 24 | 58.1 | 60.9
  Week 32 | 58.1 | 60.9
  Week 40 | 54.8 | 64.2
  Week 48 | 53.8 | 57.5
  Week 52 | 52.7 | 60.3

13. Secondary Outcome: Percentage of Participants With Clinical and Biomarker Remission at Weeks 8, 16 and 52
Description: Percentage of participants with clinical and biomarker remission was defined as the percentage of participants with CDAI <150, CRP <= 3 mg/L, and also fecal calprotectin <=250 micrograms per gram (mcg/g). The CDAI score is used to quantify the symptoms of participants with Crohn's Disease. CDAI score ranges from 0 to approximately 600; higher score indicates higher disease activities. A decrease in CDAI over time indicates improvement in disease activity.
Time Frame: At Weeks 8, 16 and 52
Population: FAS which was defined as all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab | Ustekinumab
Number analyzed (Participants) | 195 | 191
percentage of participants
  Week 8 | 19.5 | 14.1
  Week 16 | 29.7 | 18.8
  Week 52 | 27.2 | 20.9

14. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: Percentage of participants with AE were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Time Frame: Up to Week 52 and up to Week 76
Population: Safety analysis set included all the participants who were randomized and received at least one administration of study agent in the study.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab | Ustekinumab
Number analyzed (Participants) | 195 | 191
percentage of participants
  Up to Week 52 | 77.9 | 80.1
  Up to Week 76 | 80.0 | 81.7

15. Secondary Outcome: Percentage of Participants With Infections
Description: Percentage of participants with infections were reported.
Time Frame: Up to Week 52 and up to Week 76
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab | Ustekinumab
Number analyzed (Participants) | 195 | 191
percentage of participants
  Up to Week 52 | 40.5 | 34.0
  Up to Week 76 | 43.1 | 37.2

16. Secondary Outcome: Percentage of Participants With Serious Infections
Description: Percentage of participants with serious infections were reported.
Time Frame: Up to Week 52 and up to Week 76
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab | Ustekinumab
Number analyzed (Participants) | 195 | 191
percentage of participants
  Up to Week 52 | 2.6 | 2.1
  Up to Week 76 | 3.1 | 3.7

17. Secondary Outcome: Percentage of Participants With Serious Adverse Events (SAEs)
Description: Percentage of participants with SAEs were reported. A SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect and may jeopardize participant and/or may require medical or surgical intervention to prevent one of the outcomes listed above. Coronavirus disease 2019 (COVID-19) related adverse events are adverse events with any of the following preferred terms "COVID-19", "Asymptomatic COVID-19", "Suspected COVID-19", "COVID-19 pneumonia", "severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) test positive" or with a reported term containing the string "COVI.
Time Frame: Up to Week 52 and up to Week 76
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab | Ustekinumab
Number analyzed (Participants) | 195 | 191
percentage of participants
  Up to Week 52 | 16.4 | 13.1
  Up to Week 52: COVID-19 related SAEs | 0 | 0
  Up to Week 76 | 19.5 | 15.2
  Up to Week 76: COVID-19 related SAEs | 0 | 0.5

18. Secondary Outcome: Percentage of Participants With Anti-drug Antibodies
Description: Percentage of participants with anti-drug antibodies were reported. Serum samples were assessed for anti-drug antibodies. Anti-drug assays were performed for ustekinumab and adalimumab.
Time Frame: Up to Week 52
Population: Immunogenicity analysis set included all participants who had received at least 1 administration of study agent and have at least one valid blood sample drawn for detection of antibodies to study agent.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab | Ustekinumab
Number analyzed (Participants) | 195 | 190
percentage of participants | 74.4 | 2.1

ADVERSE EVENTS:
Time Frame: Up to 81 weeks
Description: Safety analysis set included all the participants who were randomized and received at least one administration of study agent in the study.
Arm/Group | Adalimumab | Ustekinumab
All-Cause Mortality (participants affected / at risk) | 1/195 | 0/191
Serious Adverse Events (participants affected / at risk) | 38/195 | 29/191
Other Adverse Events (participants affected / at risk) | 151/195 | 152/191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=195) | Ustekinumab (N=191)
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Angina Unstable (Cardiac disorders) | 0 | 1
Venolymphatic Malformation (Congenital, familial and genetic disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Anal Fistula (Gastrointestinal disorders) | 1 | 1
Crohn's Disease (Gastrointestinal disorders) | 17 | 5
Duodenal Stenosis (Gastrointestinal disorders) | 0 | 2
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Ileal Stenosis (Gastrointestinal disorders) | 1 | 2
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 2
Intestinal Perforation (Gastrointestinal disorders) | 1 | 0
Intestinal Stenosis (Gastrointestinal disorders) | 1 | 0
Intussusception (Gastrointestinal disorders) | 1 | 0
Large Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Large Intestine Perforation (Gastrointestinal disorders) | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 3
Subileus (Gastrointestinal disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 0 | 1
Sudden Death (General disorders) | 1 | 0
Bile Duct Stone (Hepatobiliary disorders) | 1 | 0
Cholecystitis Chronic (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1
Abdominal Abscess (Infections and infestations) | 0 | 1
Anal Abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 0 | 1
Clostridium Difficile Infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Epididymitis (Infections and infestations) | 0 | 1
Paracoccidioides Infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 1
Pulmonary Tuberculosis (Infections and infestations) | 1 | 0
Rectal Abscess (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1
Crush Injury (Injury, poisoning and procedural complications) | 0 | 1
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Foot Deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness Postural (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 0 | 1
Psychotic Disorder (Psychiatric disorders) | 1 | 1
Ovarian Cyst (Reproductive system and breast disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Peripheral Vascular Disorder (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=195) | Ustekinumab (N=191)
Anaemia (Blood and lymphatic system disorders) | 7 | 6
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Extrasystoles (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 2
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Syringomyelia (Congenital, familial and genetic disorders) | 1 | 0
Ear Haemorrhage (Ear and labyrinth disorders) | 0 | 1
Ear Pain (Ear and labyrinth disorders) | 1 | 0
Ear Swelling (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 4 | 7
Blepharospasm (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Choroidal Effusion (Eye disorders) | 0 | 1
Conjunctivitis Allergic (Eye disorders) | 1 | 0
Dry Eye (Eye disorders) | 1 | 2
Eye Pruritus (Eye disorders) | 0 | 1
Eyelid Cyst (Eye disorders) | 0 | 1
Eyelid Oedema (Eye disorders) | 1 | 0
Foreign Body Sensation in Eyes (Eye disorders) | 0 | 1
Glaucoma (Eye disorders) | 1 | 0
Iridocyclitis (Eye disorders) | 1 | 0
Iritis (Eye disorders) | 1 | 0
Keratitis (Eye disorders) | 1 | 0
Retinal Detachment (Eye disorders) | 1 | 0
Swelling of Eyelid (Eye disorders) | 0 | 1
Uveitis (Eye disorders) | 0 | 1
Vision Blurred (Eye disorders) | 3 | 1
Abdominal Distension (Gastrointestinal disorders) | 2 | 2
Abdominal Hernia (Gastrointestinal disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 16 | 25
Abdominal Pain Lower (Gastrointestinal disorders) | 2 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 5 | 7
Abdominal Tenderness (Gastrointestinal disorders) | 0 | 1
Anal Fissure (Gastrointestinal disorders) | 2 | 7
Anal Fistula (Gastrointestinal disorders) | 0 | 2
Anal Pruritus (Gastrointestinal disorders) | 0 | 3
Anal Stenosis (Gastrointestinal disorders) | 0 | 1
Anorectal Discomfort (Gastrointestinal disorders) | 2 | 0
Chronic Gastritis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 7 | 7
Crohn's Disease (Gastrointestinal disorders) | 29 | 20
Defaecation Urgency (Gastrointestinal disorders) | 0 | 2
Dental Caries (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 11
Diarrhoea Haemorrhagic (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 4 | 4
Enlarged Uvula (Gastrointestinal disorders) | 0 | 1
Eosinophilic Oesophagitis (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 4
Food Poisoning (Gastrointestinal disorders) | 1 | 0
Frequent Bowel Movements (Gastrointestinal disorders) | 1 | 2
Gastric Ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1
Gastritis Erosive (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 5 | 6
Gingival Swelling (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 3
Haemorrhoids (Gastrointestinal disorders) | 1 | 3
Ileal Stenosis (Gastrointestinal disorders) | 0 | 1
Large Intestinal Stenosis (Gastrointestinal disorders) | 0 | 1
Lip Blister (Gastrointestinal disorders) | 0 | 1
Mouth Haemorrhage (Gastrointestinal disorders) | 1 | 0
Mouth Ulceration (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 9 | 12
Proctitis (Gastrointestinal disorders) | 1 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 3
Rectal Tenesmus (Gastrointestinal disorders) | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 4 | 11
Asthenia (General disorders) | 0 | 1
Chest Discomfort (General disorders) | 2 | 0
Chest Pain (General disorders) | 0 | 2
Drug Intolerance (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 8
Impaired Healing (General disorders) | 1 | 0
Influenza Like Illness (General disorders) | 0 | 2
Injection Site Bruising (General disorders) | 0 | 1
Injection Site Erythema (General disorders) | 13 | 3
Injection Site Haematoma (General disorders) | 0 | 1
Injection Site Irritation (General disorders) | 1 | 0
Injection Site Oedema (General disorders) | 3 | 0
Injection Site Pain (General disorders) | 3 | 1
Injection Site Pruritus (General disorders) | 7 | 2
Injection Site Rash (General disorders) | 2 | 1
Injection Site Reaction (General disorders) | 1 | 0
Injection Site Swelling (General disorders) | 4 | 0
Malaise (General disorders) | 1 | 2
Medical Device Pain (General disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 0
Oedema Peripheral (General disorders) | 0 | 5
Pain (General disorders) | 2 | 1
Peripheral Swelling (General disorders) | 2 | 2
Pyrexia (General disorders) | 8 | 6
Suprapubic Pain (General disorders) | 1 | 0
Vessel Puncture Site Haematoma (General disorders) | 0 | 1
Cholangitis Sclerosing (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Hepatic Steatosis (Hepatobiliary disorders) | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Drug Hypersensitivity (Immune system disorders) | 1 | 0
Seasonal Allergy (Immune system disorders) | 2 | 0
Abdominal Abscess (Infections and infestations) | 0 | 2
Abscess Limb (Infections and infestations) | 0 | 1
Abscess Oral (Infections and infestations) | 1 | 0
Acute Sinusitis (Infections and infestations) | 2 | 0
Anal Abscess (Infections and infestations) | 1 | 1
Asymptomatic COVID-19 (Infections and infestations) | 2 | 2
Bacterial Vulvovaginitis (Infections and infestations) | 0 | 1
Blister Infected (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 3 | 0
Bronchitis Bacterial (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 4 | 1
Candida Infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Cervicitis (Infections and infestations) | 0 | 1
Conjunctivitis (Infections and infestations) | 2 | 0
Cystitis (Infections and infestations) | 0 | 3
Dermatophytosis of Nail (Infections and infestations) | 1 | 0
Ear Infection (Infections and infestations) | 1 | 3
Eczema Infected (Infections and infestations) | 0 | 1
Eye Infection (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 1 | 0
Fungal Skin Infection (Infections and infestations) | 1 | 0
Furuncle (Infections and infestations) | 1 | 2
Gastroenteritis (Infections and infestations) | 3 | 3
Gastroenteritis Viral (Infections and infestations) | 0 | 1
Gastrointestinal Bacterial Overgrowth (Infections and infestations) | 0 | 1
Gastrointestinal Viral Infection (Infections and infestations) | 0 | 1
Genital Herpes (Infections and infestations) | 1 | 1
Hepatitis E (Infections and infestations) | 0 | 1
Herpes Zoster (Infections and infestations) | 2 | 1
Herpes Zoster Disseminated (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 5 | 6
Large Intestine Infection (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0
Latent Tuberculosis (Infections and infestations) | 1 | 0
Localised Infection (Infections and infestations) | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 2 | 1
Nasopharyngitis (Infections and infestations) | 20 | 14
Onychomycosis (Infections and infestations) | 0 | 1
Oral Candidiasis (Infections and infestations) | 0 | 1
Oral Herpes (Infections and infestations) | 11 | 1
Oropharyngeal Candidiasis (Infections and infestations) | 0 | 1
Otitis Externa (Infections and infestations) | 1 | 0
Otitis Media (Infections and infestations) | 1 | 1
Pharyngitis (Infections and infestations) | 2 | 1
Pharyngitis Streptococcal (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 0 | 1
Post Procedural Infection (Infections and infestations) | 0 | 2
Postoperative Wound Infection (Infections and infestations) | 0 | 1
Rectal Abscess (Infections and infestations) | 0 | 2
Respiratory Syncytial Virus Infection (Infections and infestations) | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 2 | 0
Respiratory Tract Infection Viral (Infections and infestations) | 3 | 1
Rhinitis (Infections and infestations) | 3 | 2
Salmonellosis (Infections and infestations) | 1 | 0
Septic Shock (Infections and infestations) | 0 | 1
Sinobronchitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 7 | 3
Staphylococcal Skin Infection (Infections and infestations) | 1 | 0
Streptococcal Infection (Infections and infestations) | 2 | 0
Suspected COVID-19 (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 3 | 3
Tooth Abscess (Infections and infestations) | 0 | 3
Tooth Infection (Infections and infestations) | 1 | 2
Tracheobronchitis (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 15 | 13
Urinary Tract Infection (Infections and infestations) | 11 | 7
Vaginal Infection (Infections and infestations) | 0 | 1
Viral Infection (Infections and infestations) | 4 | 3
Viral Upper Respiratory Tract Infection (Infections and infestations) | 2 | 2
Vulvitis (Infections and infestations) | 0 | 1
Vulvovaginal Candidiasis (Infections and infestations) | 1 | 4
Vulvovaginal Mycotic Infection (Infections and infestations) | 1 | 2
Arthropod Bite (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 2
Exposure to Toxic Agent (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Foreign Body in Eye (Injury, poisoning and procedural complications) | 2 | 0
Hand Fracture (Injury, poisoning and procedural complications) | 1 | 1
Joint Injury (Injury, poisoning and procedural complications) | 1 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 2 | 2
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 3
Post Procedural Inflammation (Injury, poisoning and procedural complications) | 1 | 0
Procedural Anxiety (Injury, poisoning and procedural complications) | 1 | 0
Procedural Dizziness (Injury, poisoning and procedural complications) | 0 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 1 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 1
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 1
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 1
Splinter (Injury, poisoning and procedural complications) | 0 | 1
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 1
Tooth Fracture (Injury, poisoning and procedural complications) | 0 | 1
Tooth Injury (Injury, poisoning and procedural complications) | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 6 | 2
Aspartate Aminotransferase Increased (Investigations) | 3 | 3
Blood Creatinine Increased (Investigations) | 2 | 0
Blood Folate Decreased (Investigations) | 1 | 0
Blood Glucose Increased (Investigations) | 0 | 1
Blood Phosphorus Increased (Investigations) | 1 | 0
Blood Pressure Increased (Investigations) | 1 | 0
Blood Testosterone Decreased (Investigations) | 0 | 1
Body Temperature Increased (Investigations) | 0 | 1
C-Reactive Protein Increased (Investigations) | 2 | 2
Colonoscopy Abnormal (Investigations) | 0 | 1
Faecal Calprotectin Increased (Investigations) | 1 | 1
Granulocyte Count Decreased (Investigations) | 1 | 0
Haematocrit Increased (Investigations) | 1 | 0
Heart Rate Increased (Investigations) | 1 | 0
Hepatic Enzyme Increased (Investigations) | 1 | 2
Human Chorionic Gonadotropin Increased (Investigations) | 1 | 0
Liver Function Test Increased (Investigations) | 2 | 2
Mycobacterium Tuberculosis Complex Test Positive (Investigations) | 1 | 1
Transaminases Increased (Investigations) | 2 | 0
Urine Output Increased (Investigations) | 1 | 0
Vitamin B12 Decreased (Investigations) | 1 | 0
Weight Decreased (Investigations) | 3 | 0
Weight Increased (Investigations) | 0 | 2
White Blood Cell Count Decreased (Investigations) | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Folate Deficiency (Metabolism and nutrition disorders) | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 2
Hypoferritinaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Hypovitaminosis (Metabolism and nutrition disorders) | 0 | 1
Impaired Fasting Glucose (Metabolism and nutrition disorders) | 0 | 1
Iron Deficiency (Metabolism and nutrition disorders) | 0 | 1
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 1
Vitamin B12 Deficiency (Metabolism and nutrition disorders) | 0 | 3
Vitamin D Deficiency (Metabolism and nutrition disorders) | 1 | 5
Ankylosing Spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 13
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis Enteropathic (Musculoskeletal and connective tissue disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 8
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Diastasis Recti Abdominis (Musculoskeletal and connective tissue disorders) | 0 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 2 | 0
Lupus-Like Syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3 | 2
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 3
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Plantar Fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Psoriatic Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
SAPHO Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal Pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Temporomandibular Joint Syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Tenosynovitis Stenosans (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign Neoplasm of Eye (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dysplastic Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Seborrhoeic Keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Amnesia (Nervous system disorders) | 0 | 1
Cervical Radiculopathy (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 2
Dizziness Postural (Nervous system disorders) | 0 | 4
Dysgeusia (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 14 | 25
Hemiplegic Migraine (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 2 | 1
Lethargy (Nervous system disorders) | 0 | 1
Memory Impairment (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 2
Migraine with Aura (Nervous system disorders) | 1 | 0
Nerve Compression (Nervous system disorders) | 0 | 2
Paraesthesia (Nervous system disorders) | 1 | 1
Presyncope (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 3
Sinus Headache (Nervous system disorders) | 0 | 4
Syncope (Nervous system disorders) | 1 | 1
Tension Headache (Nervous system disorders) | 1 | 1
Tremor (Nervous system disorders) | 0 | 2
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Affect Lability (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 3 | 6
Anxiety Disorder (Psychiatric disorders) | 1 | 1
Depressed Mood (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 4 | 2
Insomnia (Psychiatric disorders) | 3 | 1
Panic Attack (Psychiatric disorders) | 1 | 0
Sleep Disorder (Psychiatric disorders) | 0 | 2
Stress (Psychiatric disorders) | 0 | 1
Azotaemia (Renal and urinary disorders) | 1 | 0
Chronic Kidney Disease (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 2
Haematuria (Renal and urinary disorders) | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 1
Nocturia (Renal and urinary disorders) | 0 | 1
Amenorrhoea (Reproductive system and breast disorders) | 0 | 1
Cervical Dysplasia (Reproductive system and breast disorders) | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 2 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1
Nipple Pain (Reproductive system and breast disorders) | 0 | 1
Ovarian Cyst (Reproductive system and breast disorders) | 2 | 1
Semen Discolouration (Reproductive system and breast disorders) | 0 | 1
Uterine Haemorrhage (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal Discomfort (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Asthma Late Onset (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nasal Crusting (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 | 9
Pharyngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Acne (Skin and subcutaneous tissue disorders) | 3 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 7
Brow Ptosis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 1
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 4
Drug Eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 4 | 4
Eczema Nummular (Skin and subcutaneous tissue disorders) | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 4 | 0
Erythema Nodosum (Skin and subcutaneous tissue disorders) | 1 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Ingrowing Nail (Skin and subcutaneous tissue disorders) | 0 | 1
Night Sweats (Skin and subcutaneous tissue disorders) | 2 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Post Inflammatory Pigmentation Change (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2
Pseudofolliculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 3 | 2
Rash (Skin and subcutaneous tissue disorders) | 6 | 3
Rash Erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Rash Papular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash Pruritic (Skin and subcutaneous tissue disorders) | 2 | 1
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 1
Scar Pain (Skin and subcutaneous tissue disorders) | 1 | 0
Sebaceous Hyperplasia (Skin and subcutaneous tissue disorders) | 0 | 1
Seborrhoeic Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 2 | 1
Skin Fissures (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 2
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 1
Tonsillectomy (Surgical and medical procedures) | 0 | 1
Aortic Arteriosclerosis (Vascular disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1
Flushing (Vascular disorders) | 1 | 0
Hot Flush (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 5 | 3
Raynaud's Phenomenon (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/36/NCT03464136/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/36/NCT03464136/SAP_001.pdf